CLINICAL TRIAL: NCT02405572
Title: Feeding Tolerance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 14.32.US.INF
Record Dates: First submitted 2015-02-23; First posted 2015-04-01 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: formula-fed; infants
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formula 1 (Active Comparator): infant formula
  Interventions: Other: infant formula
- Formula 2 (Active Comparator): infant formula
  Interventions: Other: infant formula

INTERVENTIONS:
Other: infant formula — infant formulas

SUMMARY:
Crossover study of 2 infant formulas

DETAILED DESCRIPTION:
Exclusively formula-fed infants will participate in two 2-week feeding periods of 2 infant formulas. Daily tolerance records will be kept by caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full-term (> 37 weeks gestation)
* 0-2 months (birth-56 days) of age on enrollment
* Infant exclusively formula-fed for at least 2 days prior to enrollment
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Known or suspected cow-milk allergy
* Congenital illness or malformation
* Significant prenatal and/or postnatal disease
* Currently participating in another clinical study

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
stool consistency | 2 weeks
  caregivers will document on diary records

SECONDARY OUTCOMES:
spit-up pattern | 2 weeks
  caregivers will document on diary records
formula intake | 2 weeks
  caregivers will document on diary records
adverse events | 2 weeks
  assessed throughout the study
stool pattern | 2 weeks
  caregivers will document on diary records
mood | 2 weeks
  caregivers will document on diary records
sleep pattern | 2 weeks
  caregivers will document on diary records

CONTACTS AND LOCATIONS:
Overall Officials: Rich Litov, PhD, Principal Investigator — Pedia Research
Locations (2):
- United States (2):
  - Pedia Research, Owensboro, Kentucky
  - Tanner Clinic, Layton, Utah